CLINICAL TRIAL: NCT05006638
Title: Assessing The Role Of Intravenous Lipid Emulsion As A Life Saving Therapy In Pesticides Toxicity: A Randomized Controlled Trial In Poison Control Center Of Ain Shams University Hospitals
Brief Title: Assessing The Role Of Intravenous Lipid Emulsion As A Life Saving Therapy In Pesticides Toxicity
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aya Sabry Mohamed Mohamed (Other)
Responsible Party: Sponsor-Investigator, Aya Sabry Mohamed Mohamed, Assistant lecturer of forensic medicine and clinical toxicology department faculty of medicine Ain shams university, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MD27/2021
Record Dates: First submitted 2021-08-08; First posted 2021-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Pesticide Poisoning
MeSH Terms: interventions — Fat Emulsions, Intravenous; Atropine; Obidoxime Chloride; Ondansetron

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): will receive the traditional supportive treatment according to (PCC-ASUH) protocol
  Interventions: Drug: Atropine; Drug: Toxogonin; Drug: Sodium Bicarbonate Powder and ondansetron
- case group (Active Comparator): will receive the traditional supportive treatment plus administration of ILE (20%) 1.5 ml/kg as a bolus over 2-3 minutes. Followed immediately by an infusion of 20 % lipid emulsion at a rate of 0.25 mL/kg/min. After 3 minutes of this infusion rate, response to the bolus and initial infusion should be assessed. If there has been a significant response, the infusion rate can be adjusted to 0.025 mL/kg/min with monitoring of blood pressure, heart rate, and other available hemodynamic parameters during the infusion with a maximum dose of 10 mL/kg
  Interventions: Drug: Lipid Emulsion, Intravenous; Drug: Atropine; Drug: Toxogonin; Drug: Sodium Bicarbonate Powder and ondansetron

INTERVENTIONS:
Drug: Lipid Emulsion, Intravenous — Lipid emulsion is a mixture of soybean oil, egg phospholipids, glycerine, and is available in 10%, 20%, and 30% strengths. It has been used for decades as parenteral nutrition and for caloric supplementation and essential fatty acid deficiency. It has also been used as a carrier for lipid soluble medications
  Arms: case group
Drug: Atropine — a drug used as an antidote for some types of pesticides
Drug: Toxogonin — a drug used as an antidote for some types of pesticides
Drug: Sodium Bicarbonate Powder and ondansetron — standard of care for treatment of aluminuim phosphide is provided for patients poisoned with aluminuim phosphide

SUMMARY:
Intravenous lipid emulsion is an established, effective treatment for local anesthetic systemic toxicity. It is also efficacious in animal models of severe cardiotoxicity caused by a number of other medications. Recent case reports of successful resuscitation suggest the efficacy of lipid emulsion infusion for treating non-local anesthetic overdoses across a wide spectrum of drugs. The present study will focus on the potential role of intravenous lipid emulsion as an adjuvant therapy in pesticides toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute pesticide intoxications with poison severity score 2 or 3 admitted in ICU of PCC-ASUH

Exclusion Criteria:

* Patients less than 18 years and more than 65 years.
* Pregnant and lactating females.
* Presence of medical diseases (e.g. renal, hepatic, cardiovascular, neurological diseases and chronic pancreatitis.)
* Allergy to soya-, egg-or peanut protein

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
mortality rate reduction | 1 year
  the primary end point is to lower the mortality rate for patients poisoned with pesticides
organ damage reduction | 1 year
  another primary end point is to reduce organ damage and injury for survivors

CONTACTS AND LOCATIONS:
Locations (1):
- Poison Control Center of Ain-Shams University hospitals, Cairo, Abbasya, Egypt